CLINICAL TRIAL: NCT06414395
Title: The Effects of Different Loading Doses of Dexmedetomidine on The Bispectral Index-Guided Propofol Sedation in Patients Undergoing Advanced Upper Gastrointestinal Endoscopic Procedures: A Randomized Control Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Sameh Mohamed Elaidy, Assistant lecturer, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PT (704)
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: GIT Endoscopy; Procedural Sedation
MeSH Terms: interventions — Dexmedetomidine; Injections

STUDY DESIGN:
Intervention Model Description: This study hypothesizes that lower doses of dexmedetomidine (0.25 µg.kg-1 or the 0.5 µg.kg-1) can co-produce adequate propofol sparing sedation that is not inferior to the standard dose of 1µg.kg-1 and without significantly prolonging the propofol recovery time or increasing the total propofol consumption.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be performed using computer generated numbers with Random Allocation Software in a 1:1:1:1 ratio. The patient's allocation and drug administration instructions will be kept in consequentially numbered opaque envelopes (equal number per each group). A colleague, not participating to the study, will be responsible for study drugs preparation & labelling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- The Dexmedetomidine Group D1 (Experimental): D1 group will receive 1µg.kg as a loading dose over 10 minutes, followed by maintenance 0.5 µg.kg.
  Interventions: Drug: Precedex (Dexmedetomidine) 200 MCG in 2 ML Injection
- The Dexmedetomidine Group D 0.5 (Experimental): D 0.5 group will receive 0.5 µg.kg as a loading dose over 10 minutes, followed by maintenance 0.5 µg.kg
  Interventions: Drug: Precedex (Dexmedetomidine) 200 MCG in 2 ML Injection
- The Dexmedetomidine Group D0.25 (Experimental): D 0.25 group will receive 0.25 µg.kg as a loading dose over 10 minutes, followed by maintenance 0.5 µg.kg
  Interventions: Drug: Precedex (Dexmedetomidine) 200 MCG in 2 ML Injection
- The Dexmedetomidine Group D 0 (Placebo Comparator): D 0 group will receive a placebo saline infusion over 10 minutes and then will receive 50 ml of normal saline as a placebo
  Interventions: Other: C group: Patients received saline infusion over 10 minutes

INTERVENTIONS:
Drug: Precedex (Dexmedetomidine) 200 MCG in 2 ML Injection — The Effects of Different Loading Doses of Dexmedetomidine on The Bispectral Index-Guided Propofol Sedation in Patients Undergoing Advanced Upper Gastrointestinal Endoscopic Procedures: A Randomized Control Study
  Arms: The Dexmedetomidine Group D 0.5; The Dexmedetomidine Group D0.25; The Dexmedetomidine Group D1
Other: C group: Patients received saline infusion over 10 minutes — the group will receive normal saline infusion over 10 minutes.
  Other Names: Placebo
  Arms: The Dexmedetomidine Group D 0

SUMMARY:
Propofol is currently the most common drug used but has drawbacks like narrow therapeutic window and potential complications.

Dexmedetomidine is an attractive alternative due to its unique properties like minimal respiratory depression.

Studies are ongoing to find the optimal use of dexmedetomidine for these procedures. A combination of propofol and dexmedetomidine might be ideal, but the best balance between the two drugs needs further investigation.

DETAILED DESCRIPTION:
Advanced upper gastrointestinal tract procedures such as Endoscopic retrograde cholangiopancreatography (ERCP) & Endoscopic ultrasound (EUS) are very important diagnostic and therapeutic procedures for the diagnosis & management of many pancreatobiliary pathologies whether benign or malignant (1-4). These procedures require moderate-deep sedation with the patient lying in the lateral or semi-prone position to provide the operator easier access & insertion while permitting fluoroscopic visualisation (1-4).

Propofol sedation is currently the most popular drug used for advanced endoscopic procedures because of its shorter half-life which results in a shorter recovery time than conventional sedation (benzodiazepine &/or opioid) (5). Propofol was administered initially by intermittent boluses but later on was superseded by continuous infusion guided by clinical scoring, e.g., Ramsey sedation score (6), by target-controlled infusion (TCI) (7) or more recently by bispectral index (BIS) monitoring (8).

Propofol, however, has a narrow therapeutic window that may cause fluctuation of the level of sedation from moderately deep sedation to near general anesthesia. Not only that but also propofol sedation is associated with many other complications including apnoea, airway obstruction desaturation, hypotension, bradycardia, gagging, restlessness, regurgitation & vomiting & delayed recovery (9).

Dexmedetomidine, a highly specific, potent and selective α2-adrenoceptor agonist, was originally introduced as a sedative for critically ill mechanically ventilated patients [9]. In addition to sedation, it has a group of unique properties in the form of analgesia, reduction of sympathetic tone and attenuation of the neuroendocrine and hemodynamic responses to anesthesia and surgery with minimal respiratory depression, making it an attractive agent for perioperative sedation especially in remote areas outside the operating theatres (6,10).

The quest to replace propofol coupled with the unique sedo-analgesic properties of dexmedetomidine resulted in the interest in the use of dexmedetomidine for providing sedation for advanced endoscopic procedure (6,10).

In 2021, Srivastava et al (6), studied the effects dexmedetomidine as a sole sedative agent in the form of a loading dose of 1 µg.kg-1 followed by 0.5 µg.kg-1.hr-1 continuous infusion. They reported that although this dexmedetomidine regimen produced adequate sedation in many patients yet it was associated with a relatively high sedation failure rate requiring rescue propofol boluses (6). Moreover, dexmedetomidine was associated with bradycardia & hypotension (6,7,11).

It was 2013, When Wang et al (12), examined the propofol sparing effect of various dexmedetomidine loading doses ranging between 0.25 & 1 µg.kg-1 followed by a fixed infusion of 0.5 µg.kg-1.hr-1 and reported a dose dependent reduction of propofol requirements for induction of sedation (12). However, they did not investigate the impact of these dexmedetomidine doses on the total propofol consumption for the whole procedure, the incidence of adverse events or the recovery profile of such a combination in the context of sedation for advanced endoscopic procedures. Thus, the" sweet spot" (13), where there is a maximal synergism between propofol and dexmedetomidine, is still to be identified.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65
* Both sexes
* ASA I-II
* BMI <35

Exclusion Criteria:

* Patients' refusal to participate
* ASA III-IV
* BMI > 35
* Patients who are considered high aspiration risk, e.g., gastric outlet obstruction
* Allergy to any medications used
* Diabetics
* Any patient receiving cardioactive drugs, e.g., Beta blockers, Calcium channel blockers, Inhaled B2 bronchodilators)
* Patients with Pacemakers or heart rate below 50 beat/min
* Pregnant women
* Habitual Drug abusers
* Patients who had to be intubated during the procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
• Recovery time of each group: the time from ending the infusions till a modified Aldrete score (MAS) score of ≥ 9 is reached. | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz Research Institute, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided